CLINICAL TRIAL: NCT01116401
Title: Impact of Experimentally Induced Hot Flashes on Sleep and Mood Disturbance
Brief Title: Impact of Hot Flashes on Sleep and Mood Disturbance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Hadine Joffe, MD, Vice Chair for Psychiatry Research, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2009-P-001557; 5R01MH082922 (NIH)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Menopause; Depression; Hot Flashes
Keywords: Hot Flashes; Sleep disturbance; Lupron; Menopause
MeSH Terms: conditions — Depression; Hot Flashes; Parasomnias | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GnRH Agonist Injection (Experimental): We will be administering an injection of leuprolide acetate (a GnRH agonist) to all participants.
  Interventions: Drug: leuprolide

INTERVENTIONS:
Drug: leuprolide — Leuprolide acetate is a widely used GnRH agonist. In this protocol, leuprolide will be administered at a dose routinely used for treatment of endometriosis and uterine fibroids in women (one 3.75-mg intramuscular injection).
  Other Names: Lupron

SUMMARY:
We plan to enroll premenopausal women in a trial investigating the impact of hot flashes developed in response to an injection of a gonadotropin-releasing hormone agonist (GnRHa), leuprolide (brand name: Lupron), on sleep disruption and mood. This study is designed to mimic the menopause transition. We will collect data on sleep disruption and mood changes to assess their relationship to the development of hot flashes.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years old
* Premenopausal
* Willingness to use barrier methods of contraception during study and after completion of study until menses resume
* Good general health

Exclusion Criteria:

* Pregnancy or currently breastfeeding
* Hot flushes
* Mid-luteal phase progesterone <3ng/mL
* Clinically significant abnormalities in screening blood tests
* BMI > 35 kg/m2
* Previously diagnosed osteoporosis or osteopenia
* Clinically significant depressive symptoms
* Psychiatric illness
* Sleep apnea or periodic limb movement of sleep (PLMS)
* Contraindication, hypersensitivity, or previous allergic reaction to GnRH agonists
* Current or recent use of centrally active medications
* Current or recent use of systemic hormone medications
* Night shift workers
* Current use of over-the-counter (OTC) medications that may affect hot flashes, sleep, or mood
* Abnormal vaginal bleeding
* History of any medical diseases that may put subject at risk when treated with study medication.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2009-11-03 (Actual); Primary Completion 2011-12-29 (Actual); Study Completion 2012-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Joffe H, Crawford SL, Freeman MP, White DP, Bianchi MT, Kim S, Economou N, Camuso J, Hall JE, Cohen LS. Independent Contributions of Nocturnal Hot Flashes and Sleep Disturbance to Depression in Estrogen-Deprived Women. J Clin Endocrinol Metab. 2016 Oct;101(10):3847-3855. doi: 10.1210/jc.2016-2348. Epub 2016 Sep 28. PMID 27680875
- [Derived] Bianchi MT, Kim S, Galvan T, White DP, Joffe H. Nocturnal Hot Flashes: Relationship to Objective Awakenings and Sleep Stage Transitions. J Clin Sleep Med. 2016 Jul 15;12(7):1003-9. doi: 10.5664/jcsm.5936. PMID 26951410
- [Derived] Joffe H, Crawford S, Economou N, Kim S, Regan S, Hall JE, White D. A gonadotropin-releasing hormone agonist model demonstrates that nocturnal hot flashes interrupt objective sleep. Sleep. 2013 Dec 1;36(12):1977-85. doi: 10.5665/sleep.3244. PMID 24293774

RESULTS

PARTICIPANT FLOW:
Groups:
- GnRH Agonist Injection: One 3.75-mg intramuscular injection of leuprolide acetate
Period: Overall Study
Arm/Group | GnRH Agonist Injection
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GnRH Agonist Injection
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Wake After Sleep Onset (WASO)
Description: Wake after sleep onset (WASO) is calculated by averaging the number of minutes spent awake after initiating sleep each night from the two ambulatory polysomnography studies conducted at baseline and the two ambulatory polysomnography studies conducted four weeks after the GnRHa injection.
Time Frame: baseline and 4 weeks
Measure: Number (95% Confidence Interval); unit: percent change
Arm/Group | GnRH Agonist Injection
Number analyzed (Participants) | 29
percent change | 62 [18 to 106]
Statistical Analysis 1: Comparison: GnRH Agonist Injection; Test type: Superiority or Other; p = 0.007, Regression, Linear

2. Secondary Outcome: Change in Montgomery-Asperg Depression Rating Scale (MADRS)
Description: The Montgomery-Åsberg Depression Rating Scale is a widely used 10-item clinician-rated scale that describes the severity of depressive symptoms. It has a range of 0-60 with higher scores indicating greater symptom burden. Participants were assessed at baseline and four weeks after the GnRHa injection in order to calculate the change in MADRS score.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GnRH Agonist Injection
Number analyzed (Participants) | 29
units on a scale | 3.1 (5.4)
Statistical Analysis 1: Comparison: GnRH Agonist Injection; Test type: Superiority or Other; p < 0.01, Regression, Linear

ADVERSE EVENTS:
Description: To measure hot flashes, all subjects completed daily hot flash diaries through the fourth week after receiving the GnRHa and completing both ambulatory posttreatment PSGs. Nighttime hot flashes were measured objectively using an ambulatory skin conductance monitor concurrent with both post-treatment polysomnographic assessments.
Arm/Group | GnRH Agonist Injection
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 28/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GnRH Agonist Injection (N=29)
Hot flashes (Blood and lymphatic system disorders) | 25
Headache/migraine (Nervous system disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 3
Decreased Sleep/Insomnia (Nervous system disorders) | 4
Irritability/Mood changes (Psychiatric disorders) | 7
Spotting (Reproductive system and breast disorders) | 12
Heavy menstrual bleeding (Reproductive system and breast disorders) | 3
Abdominal cramps (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes